CLINICAL TRIAL: NCT06615362
Title: Autogenous Dentin Derived Barrier Membrane Versus Collagen Membrane for Guided Bone Regeneration in Immediate Implant
Brief Title: Autogenous Dentin Derived Barrier Membrane Versus Collagen Membrane
Acronym: DDBM dental
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mansoura University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: A04010222
Record Dates: First submitted 2024-09-07; First posted 2024-09-26 (Actual); Last update posted 2024-09-26 (Actual); Status verified 2024-09

CONDITIONS: TOOTH EXTRACTION; IMMEDIATE IMPLANT

STUDY DESIGN:
Intervention Model Description: Two arms: one arm Autogenous Dentin Derived Barrier Membrane ,second arm Collagen Membrane .
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Autogenous Dentin Derived Barrier Membrane (Experimental): Autogenous Dentin Derived Barrier Membrane + Xenogeneic bone graft material+ immediate implant
  Interventions: Procedure: preparation of dentin membrane from hopeless tooth for Guided Bone Regeneration in Immediate Implant
- Collagen Membrane (Experimental): Collagen Membrane + Xenogeneic bone graft material + immediate implant
  Interventions: Procedure: Collagen Membrane for Guided Bone Regeneration in Immediate Implant

INTERVENTIONS:
Procedure: preparation of dentin membrane from hopeless tooth for Guided Bone Regeneration in Immediate Implant — tooth extraction , preparation of dentin membrane ,immediate implantation ,Xenogeneic bone graft material, application of dentin derived barrier membrane
  Arms: Autogenous Dentin Derived Barrier Membrane
Procedure: Collagen Membrane for Guided Bone Regeneration in Immediate Implant — like group one but with application of collagen membrane
  Arms: Collagen Membrane

SUMMARY:
Autogenous Dentin Derived Barrier Membrane versus Collagen Membrane

DETAILED DESCRIPTION:
Autogenous Dentin Derived Barrier Membrane versus Collagen Membrane for Guided Bone Regeneration in Immediate Implant

ELIGIBILITY:
Inclusion Criteria:

1. Patient's age ranges from 18-50 years.
2. Adequate inter-arch relation and inter-occlusal space that could accommodate the implant abutment and the future restoration
3. Non-restorable tooth that needs dental extraction & guided bone regeneration for immediate implant.
4. Presence of alveolar bone defect with vertical loss of buccal bone more than a third implant thread.
5. Co-operative patients willing to complete the follow-up periods.

Exclusion Criteria:

1. Any pathological condition at site of surgery.
2. Patients with systemic diseases that contra-indicate the surgical procedure.
3. Heavy smoking.
4. Parafunctional habits such as bruxism and clenching.
5. Pregnant patients. -

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2022-04-10 (Actual); Primary Completion 2024-04-10 (Actual); Study Completion 2024-10-10 (Estimated)

PRIMARY OUTCOMES:
All patients were evaluated radiographically immediately postoperative,and after 12 months | 1 year
  Radiographic Evaluation Cone Beam Computed Tomography scan was taken to measure Marginal Bone loss and Relative bone density

CONTACTS AND LOCATIONS:
Overall Officials: Heba Elsheikh Assistant professor, Assistant professor, Study Chair — Mansoura University, faculty of dentistry ,Department of Oral and Maxillofacial
Locations (2):
- Egypt (2):
  - Mansoura University, faculty of dentistry ,Department of Oral and Maxillofacial, Al Mansurah, Eygpt
  - Elhussein Farag, Al Mansurah, Eygpt

REFERENCES:
- [Derived] Mohamad EHFA, Awad S, Abbas MH, Elsheikh HA. Autogenous dentin-derived membrane as a biologic alternative to collagen membrane for guided bone regeneration in immediate implant placement in the posterior mandible: a randomized clinical trial. Odontology. 2025 Dec 10. doi: 10.1007/s10266-025-01271-6. Online ahead of print. PMID 41372516